CLINICAL TRIAL: NCT00726336
Title: A Phase I, Open Label, Single Sequence,Drug Interaction Study Evaluating Plasma GSK1349572 and Tenofovir Pharmacokinetics in Healthy Adult Subjects (ING111604)
Brief Title: GSK1349572 Drug Interaction With Tenofovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 111604
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: healthy volunteer; pharmacokinetics; GSK1349572; integrase
MeSH Terms: interventions — dolutegravir; Tenofovir

INTERVENTIONS:
Drug: GSK1349572 and tenofovir

SUMMARY:
A study in healthy volunteers to determine whether there is a drug interaction between GSK1349572 and tenofovir

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

  * Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or
  * Is post-menopausal defined as 12 months of spontaneous amenorrhea.
* A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory. - Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt, HRT should be discontinued for 2 weeks and then the subject rescreened, as HRT can suppress FSH.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m² (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* For subjects who have received antiretroviral treatment in the past, adequate treatment options to construct HIV therapy with at least 3 active antiretrovirals for future treatment, based on review and agreement by the Investigator and the GSK Medical Monitor.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen.
* A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as:

  · An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. - Subjects with a history of cholecystectomy should be excluded.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatic diseases.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* Serum creatinine values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* ECG criteria outside protocol limits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 steady-state AUC(0-tau), Cmax and Ctau following administration of GSK1349572 50 mg q24h for 5 days and following co-administration with TDF 300 mg q24h for 5 days

SECONDARY OUTCOMES:
Plasma tenofovir steady-state AUC(0-24), Cmax and Ct following administration of TDF 300 mg q24h for 7 days alone and following co-administration with GSK1349572 50 mg q24h for 5 days.
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States